CLINICAL TRIAL: NCT02277912
Title: Efficacy of Navigated Repetitive Transcranial Magnetic Stimulation in Treatment of Central Post Stroke Pain
Brief Title: Efficacy of Transcranial Magnetic Stimulation (TMS) in Central Post Stroke Pain ( CPSP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Juhani Ojala, MD, Helsinki University Central Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: TYH2013311
Record Dates: First submitted 2014-10-22; First posted 2014-10-29 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Central Post Stroke Pain
Keywords: ICH; Stroke; Navigated; Placebo; TMS
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Transcranial Magnetic Stimulation I (Experimental): Intervention: Repetitive navigated Transcranial Magnetic Stimulation of the motor cortex
  Interventions: Device: navigated rTMS of motor cortex
- Transcranial Magnetic Stimulation II (Experimental): Intervention: Repetitive navigated Transcranial Magnetic Stimulation of the secondary somatosensory cortex
  Interventions: Device: navigated rTMS of somatosensory cortex 2
- Sham Stimulation (Sham Comparator): Intervention: Repetitive sham Transcranial Magnetic Stimulation with SHAM block of the motor cortex
  Interventions: Device: SHAM rTMS with SHAM block

INTERVENTIONS:
Device: navigated rTMS of motor cortex — Navigated repetitive transcranial magnetic stimulation of the motor cortex ( 10 Hz ) ,5 daily sessions per week for two weeks.
  Other Names: Navigated; rTMS
  Arms: Transcranial Magnetic Stimulation I
Device: navigated rTMS of somatosensory cortex 2 — Navigated repetitive transcranial magnetic stimulation of the secondary somatosensory cortex ( 10 Hz ), 5 daily sessions per week for two weeks
  Other Names: Navigated; rTMS
  Arms: Transcranial Magnetic Stimulation II
Device: SHAM rTMS with SHAM block — Repetitive SHAM transcranial magnetic stimulation of the motor cortex ( 10Hz) 5 daily sessions per week for two weeks.
  Other Names: Navigated; rTMS; Placebo
  Arms: Sham Stimulation

SUMMARY:
The aim of the study is to evaluate the analgesic effects of navigated repetitive transcranial magnetic stimulation in central post stroke pain. MRI based navigation is used to determine the exact locations for stimulation.

DETAILED DESCRIPTION:
Central post stroke pain is often very resistant to treatment. TMS has been shown to be a promising tool in treating difficult pain conditions. The best sites for stimulation are still not known and navigation has been used only in few studies.

The aim is to evaluate the analgesic effects of Navigated Repetitive Transcranial Magnetic Stimulation ( nrTMS ) on pain in a three armed crossover study. The navigation is done by using magnetic resonance imaging and stereotactic camera system. The three arms include stimulation to M1, S2 and sham stimulation to M1. 10 Hz repetitive stimulation is given to a specified location once a day 5 days a week for two weeks in each of the three arms. A months washout period is kept between each arm of the study.

Pain and other variables are followed before, during and after the study for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* MRI defined brain infarction or hemorrhage before or at the age of 65 years
* CPSP diagnostic criteria is met (definite), verified by a neurologist
* Stable analgesic medication
* Average pain NRS 4 or more

Exclusion Criteria:

* Epilepsy
* Difficult aphasia
* Dementia
* Contraindication for TMS or MRI
* Alcohol and/or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-05; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in average pain compared to baseline | 1 month after each arm of the study
  Patients will keep a pain diary for one week before stimulation and for two weeks after the stimulation. A nurse will call the patient one month after the last stimulation.

SECONDARY OUTCOMES:
Quality of life (EQ-5D) | One week after each arm of the study and 6 months after the last one
  Questionnaire EQ-5D
Depression | One week after each arm of the study and 6 months after the last stimulation
  Questionnaire
Change in average pain compared to baseline | 2,3,4,5 and 6 months after the last stimulation
  Phone call ( Numeric Rating Scale (NRS) in rest and movement )
Magnetoencephalography (MEG) | One week before and after each arms stimulations
  Changes in the irritability of the motor cortex and somatosensory cortex
Number of patients with adverse effects | From the start to the end of the study, on average 12 months per patient.
  Adverse effects are followed actively
Hands´ motor function and dexterity | One week before and after each arm of the study
  Nine hole peg, Pinch and Jamar
Cold water test | One week before and after each arm of the study
  Conditioned pain modulation (CPM)
Genetics | No time frame, just a blood sample
  Evaluation of genetical properties in terms of TMS related pain reduction

CONTACTS AND LOCATIONS:
Overall Officials: Eija Kalso, PhD, Prof., Principal Investigator — Professor of Pain Research and Management, University of Helsinki. Director of the Multidisciplinary Pain Clinic, Department of Anaesthesia and Intensive Care Medicine Helsinki University Central Hospital; Jyrki Mäkelä, MD, PhD, Study Chair — Head of laboratory, BioMag, Helsinki University Central Hospital; Erika Kirveskari, MD, PhD, Study Chair — Head and Chief Physician of Clinical Neurophysiology at Medical Imaging Center, Helsinki University Hospital

IPD SHARING:
Plan to Share IPD: No
That is not allowed according to the ethical committees decision.